CLINICAL TRIAL: NCT00014820
Title: Occupation and Asthma in an Urban Low Income Population
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 7953; R01HL062621 (NIH)
Record Dates: First submitted 2001-04-11; First posted 2001-04-12 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Patients with a diagnosis of asthma (new) (Cases): Patients with a physician diagnosis of asthma during the 7.5 years being studied who were working at the time of diagnosis, as determined by patient interviews.
- Patients with a diagnosis other than asthma (Controls): Patients (age-matched to a case patient) with a physician diagnosis other than asthma who were working at the time of diagnosis.
- Patients with a diagnosis of asthma (previous): Patients with a physician diagnosis of asthma prior to the 7.5 years being studied

SUMMARY:
To study work-related asthma in a low-income, urban population.

DETAILED DESCRIPTION:
BACKGROUND:

Work-related asthma is asthma that is attributable to, or is made worse by, environmental exposures in the workplace. Published estimates of the proportion of adult asthma attributable to occupational factors have varied widely, depending on population, methodology, and definitions, from 2 percent to 33 percent. Occupational asthma is of great public health importance because it is potentially preventable, can cause substantial disability, and in some cases is completely curable. Among adults in the United States, asthma has become a major public health problem, with rates most elevated among low income, urban, African American and Latino sectors of the population, and with substantial evidence suggesting potential occupational contributions to the excess rates. These important sectors of the U.S. population have, however, been inadequately represented in the occupational asthma research literature.

DESIGN NARRATIVE:

This was a case control study of physician-diagnosed asthma, occupation, industry, and workplace environmental exposures designed to evaluate the hypothesis that a substantial component of the asthma burden in a low income, urban, largely minority population was due to occupational factors. The study design addressed a variety of methodologic challenges including healthy worker effects, difficulty contacting and recruiting this potentially high risk population, large numbers of potential etiologic agents, mixed exposures, small workplaces, and low absolute incidence of occupational asthma.

The study population was the catchment population of Bellevue Hospital, a general hospital in lower Manhattan, New York City, with busy ambulatory care services that serve low income working communities. Cases and controls were recruited from among outpatients and inpatients at Bellevue Hospital and interviewed face-to-face or by telephone. Occupation, industry, and occupational exposures were determined by questionnaire supplemented by a Job Exposure Matrix. Odds ratios (ORs) of association between asthma and specific industrial, occupational, and exposure categories, controlled for major confounders, were estimated. The ORs were used to calculate occupation- and industry-specific Attributable Fractions, and an overall Population Attributable Fraction of asthma attributable to occupational factors. New onset occupational asthma and work-aggravated asthma were investigated separately.

ELIGIBILITY:
Exclusion criteria:

1. Subject unwilling to be interviewed or does not give informed consent
2. For nonsmokers, age under 18 or over 65. For smokers, age under 18 or over 45
3. For cases, asthma diagnosis (at Bellevue or elsewhere) prior to beginning of study period. For controls, asthma diagnosis ever.
4. Unemployed at case onset age
5. Fee-coded as Medicaid for all visits during study period
6. Fluency in either English or Spanish inadequate to communicate clearly with interviewer, or need for interpreter in language other than Spanish noted in chart
7. Medical records not HIV disease, STD, addiction-related diagnosis, or other "sensitive" diagnosis (to avoid problems of confidentiality)
8. Clear understanding of what is being asked is lacking, in judgement of interviewer
9. Responses to initial interview questions appear grossly unreliable, in the judgement of the interviewer
10. Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Bellevue Hospital who were given a diagnosis between the dates of 1/1/1996 and 6/30/2003.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2001-03; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Friedman-Jimenez, Principal Investigator — NYU Langone Health